CLINICAL TRIAL: NCT01373606
Title: An Exploratory Study of FE999908 in Patients With Hepatorenal Syndrome Type 1
Brief Title: A Study of Terlipressin in Patients With Hepatorenal Syndrome Type 1
Acronym: HRS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE999908 CS01
Record Dates: First submitted 2011-06-10; First posted 2011-06-15 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hepatorenal Syndrome Type 1
MeSH Terms: interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Terlipressin (Experimental)
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin

SUMMARY:
This is an open-label, multi-center study, investigating the efficacy and safety of terlipressin in Japanese patients with hepatorenal syndrome type 1.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were diagnosed with HRS type 1 according to the diagnostic criteria of HRS and whose serum creatinine value (SCr) doubled at 2.5 mg/dL or greater within 2 weeks or whose 24h creatinine clearance (Ccr) decreased by half at less than 20 mL/min.

Patients should meet all the following 5 criteria:

[Modified International Ascites Club's Diagnostic criteria of HRS]

1. Chronic or acute liver disease with advanced hepatic failure and portal hypertension.
2. Low glomerular filtration rate (SCr >1.5 mg/dL or 24h Ccr <40 mL/min)
3. Absence of shock, ongoing bacterial infection, current or recent (within 2 weeks) treatment with nephrotoxic drug
4. No sustained improvement in renal function (decrease in SCr to 1.5 mg/dL or less or increase in 24h Ccr to 40 mL/min or more) following diuretic withdrawal and expansion of plasma volume with 1,500 mL/24h of isotonic saline for 24 to 48h.
5. Protein urea <500 mg/dL, and no ultrasonographic evidence of obstructive uropathy or parenchymal renal disease

   * Age; 20 to 79 years

Exclusion Criteria:

* Cr value ≥5 mg/dL
* Child-Pugh Score ≥14
* Fulminant hepatitis
* Septic shock
* Hepatocellular carcinoma that does not meet the Milan Criteria
* Acute renal failure caused by contrast medium
* Chronic renal failure
* Bradycardia (heart rate <50/min)
* Hyponatraemia (serum Na <120 mEq/L)
* Ischemic heart diseases (angina pectoris, myocardial infarction), heart failure or clinically relevant arrhythmia
* Poor-controlled hypertension
* Arteriosclerosis obliterans or peripheral vascular disorder
* Cerebrovascular disorder
* Respiratory diseases such as chronic obstructive pulmonary disease
* Pregnant or possibly pregnant women and patients who or whose partner desire -pregnancy during the study period
* Patients considered by the investigator or sub-investigator as unsuitable to participate in the study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in SCr value from baseline to end of treatment | 16 days

SECONDARY OUTCOMES:
Incidence of adverse events and its severity | Up to 84 days
Laboratory test values | Up to 84 days
Vital signs | 16 days
ECG | Day 1,4,7,10,13,16
The percentage of patients with Hepatorenal syndrome reversal (SCr value <=1.5 mg/dL) | 16 days
The percentage of patients showing 20% or more reduction in SCr value from the baseline | 16 days
24h Ccr, urine volume, urea nitrogen (BUN), urinary sodium excretions | 16 days
Mean arterial blood pressure, serum Na, serum K, plasma renin activity, aldosterone, norepinephrine, antidiuretic hormone (ADH), atrial natriuresis peptide (ANP) | 16 days
Overall survival | Up to 84 days
Pharmacokinetics - assessment of blood concentration | Blood PK sample collection: pre-dose, 5, 15, 30, 60, 90, 120, 150, 180, 240, and 360 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (2):
- Japan (2):
  - Investigational site, Kansai
  - Investigational site, Kanto

REFERENCES:
- [Background] Narahara Y, Kanazawa H, Sakamoto C, Maruyama H, Yokosuka O, Mochida S, Uemura M, Fukui H, Sumino Y, Matsuzaki Y, Masaki N, Kokubu S, Okita K. The efficacy and safety of terlipressin and albumin in patients with type 1 hepatorenal syndrome: a multicenter, open-label, explorative study. J Gastroenterol. 2012 Mar;47(3):313-20. doi: 10.1007/s00535-011-0485-8. Epub 2011 Oct 25. PMID 22038555